CLINICAL TRIAL: NCT05332327
Title: Comparison of the Accuracy of Different Periodontal Probes for Peri-implant Pocket Registration
Status: Completed | Type: Observational
Sponsor: Malmö University (Other)
Responsible Party: Principal Investigator, Kristina Bertl, Principal Investigator, Malmö University
Other Study IDs: 2020-01019/2
Record Dates: First submitted 2022-04-11; First posted 2022-04-18 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Peri-Implantitis; Peri-implant Mucositis
MeSH Terms: conditions — Peri-Implantitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Various types of periodontal probes (e.g., metal probes, plastic/bendable probes, electronic periodontal probes) are used for peri-implant pocket depth registration; however, depending on the shape and size of the prosthetic restoration an accurate peri-implant pocket registration might be impeded with standard metal probes. There is currently no systematic assessment of which probe is more accurate in peri-implant pocket registration. Therefore, peri-implant pocket registration of 50 patients with a screw-retained prosthetic restoration will be recorded with 3 different periodontal probes; i.e., with a metal probe, with a plastic probe, and with an automatic periodontal probe, before and after removal of the prosthetic restoration.

ELIGIBILITY:
Inclusion Criteria:

* screw-retained prosthetic implant restoration

Exclusion Criteria:

- cemented prosthetic implant restoration

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: In 50 patients with a screw-retained prosthetic restoration the peri-implant pocket registration will be recorded with 3 different types of periodontal probes; measurements will be performed in patients for baseline assessment (i.e., before surgical intervention) as well as in patients for annual post-operative controls to include a wide range of shallow, average, and deeper peri-implant pocket depths.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2020-09-08 (Actual); Primary Completion 2023-02-13 (Actual); Study Completion 2023-02-13 (Actual)

PRIMARY OUTCOMES:
peri-implant probing pocket depth | 1 day (single measurement)
  peri-implant probing pocket depth in mm

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Periodontology, Malmö University, Malmo, Sweden